CLINICAL TRIAL: NCT07300527
Title: Cognitive Behavior Therapy for Dysfunctional Cognitive and Behavioral Patterns and Functional Outcomes Among Patients With Major Depressive Disorder-Multiples Episodes: Randomized Control Trial.
Brief Title: Cognitive Behavior Therapy Among Patients With Major Depressive Disorder-Multiple Episodes.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Government College University Faisalabad (Other)
Responsible Party: Principal Investigator, Qasir Abbas, Assistant Professor - Clinical Psychology, Government College University Faisalabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GCUF_PsychThesisTrial
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-10

CONDITIONS: Patients With Major Depressive Disorder
Keywords: patient health questionnaire,; mental help seeking attitude; motivational attitude toward changing health; digit span; GAD; Brief Quality of Life
MeSH Terms: interventions — Cognitive Behavioral Therapy; Therapeutics; Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized control trial design would be used in this study. It would be two arm study and there would be two groups an experimental and wait-list control group. Experimental group will receive intervention and control group will take treatment as usual. In this research, parallel group design would be used. We will give treatment to all participants in a parallel way. Allocation ratio and framework would be equivalence i.e., treatment group and control group would be equal number of participants. In order to collect the sample for the desired study, purposive sampling technique would be used. Patient's age range would be between 18 to 50 years. Participant would be divided into two groups. In group one, the diagnosed patients of MDD who will receive Cognitive behavior therapy would be taken 8-10 sessions. The control group will receive treatment as usual. Each of the group will be comprised of n= 40.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1st Arm (1- Experimental) (Experimental): Patients will receive cognitive behavioral Therapy
  Interventions: Behavioral: Cognitive Behavior Therapy; Drug: treatment as usual (TAU) (Control Group)
- 2nd Arm (Waitlist Control Condition) (Active Comparator): This group will receive treatment as usual
  Interventions: Drug: treatment as usual (TAU) (Control Group)

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy — This involves 10 sessions, 2 sessions per week will be conduct, session 1 ( psychoeducation about the problem, second will be cognitive Distortions, thirdly, automatic Thoughts , ABC Worksheet (Antecedent-Belief-Consequence), (Greenberger & Padesky, 2016) Daily Thought Monitoring Sheet, "Catch It - Check It - Change It" model. fourthly, Core beliefs And Dysfunctional Schemas, Downward Arrow Technique (Beck, 2011) Flashcards for Positive Beliefs, "What does that say about me?" , REFRAMING (Beck, 2011), fifth, Behavioral Activation, Increase engagement in pleasurable and meaningful activities. sixth, Memory and concentration, Enhance mindfulness and address cognitive memory concerns. To help patient focus on present moment. seventh, stress management Training, eighthly, problem solving skills, Relationship management skills, lastly, relapse Prevention, review skills, plan for future, reinforce independence.
  each session have specific goals and outcomes.
  Arms: 1st Arm (1- Experimental)
Drug: treatment as usual (TAU) (Control Group) — Participants in this arm will receive Treatment as Usual (TAU) provided by the hospital, which may include routine psychiatric care, medication management, and supportive counseling as prescribed by the treating psychiatrist. No structured psychotherapy sessions, such as CBT, will be administered during the study period. This group will serve as the control condition to compare the effects of Cognitive Behavioral Therapy (CBT) on depressive symptoms and related psychological outcomes. Standard care procedures will continue throughout the study, and participants will be assessed at the same pre- and post-intervention time points as the experimental group.

SUMMARY:
The main purpose of this study to teach the patients how to manage their depression, generalized Anxiety symptoms, mental health seeking attitude, motivation and attitude toward changing health, to improve the quality of life, and meta memory and meta cognitive functioning after using Adapted CBT. Enhance emotional regulation by helping patients identify and modify maladaptive emotional responses, thereby reducing emotional reactivity and promoting healthier coping strategies. Strengthen relapse prevention skills by equipping patients with long-term cognitive and behavioral techniques to recognize early warning signs and apply learned strategies proactively to prevent future episodes. This research would be helpful for patients etc.

DETAILED DESCRIPTION:
In this experimental study, 120 patients will be screened for eligibility from various government and private hospitals. Participants meeting the DSM-5-TR criteria for Major Depressive Disorder (multiple episodes) will be considered. Eighty eligible participants will be randomly assigned to the experimental group (n = 40) and control group (n = 40). Participants aged 18-50 years will be included. Following approval from the university and formal permissions from hospitals and patients, all ethical guidelines will be strictly observed. Eligible participants will be selected based on the inclusion criteria. The CBT group will receive two sessions per week, gradually reduced over time, with each session lasting 45-60 minutes. Pre- and post-assessments will be conducted using standardized measures to evaluate changes in depression severity and related psychological variables.

Expected outcome: The intervention is expected to significantly reduce symptoms of depression and anxiety among participants. Improvements are anticipated in help-seeking attitudes, motivation toward health behavior change, and overall quality of life. CBT is also expected to enhance meta-memory and meta-cognitive functioning. These outcomes will support the effectiveness of CBT in treating patients with recurrent MDD.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18-50 years No physical, psychiatric, or psychological conditions. patients who meet multiple Episodes. who meet DSM 5 TR Major Depressive Disorder Criteria. patients who meet moderate severity at patient health questionnaire scale .

Exclusion Criteria:

* age range: below 18 and above 50 years. presence of any physical, psychiatric, or psychological conditions. who do not meet DSM 5 TR Major Depressive Disorder Criteria. range at patient health questionnaire scale is mild , minimal or severe or moderately severe.

Ages: 18 Weeks to 50 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire PHQ-9 (Kroenke, and colleagues, 1999) | at pre-Assessment, after 5 weeks at post-Assessment
  Kroenke, and colleagues (1999) from Columbia University developed Patient Health Questionnaire. In the current study Patient Health Questionnaire 9 item questionnaire translated by (Ahmad, Hussain, Akhtar & Shah, 2018). Each item could be responded to using a 4-point Not at all = 0; several days = 1; More than half the days = 2; nearly every day = 3. The PHQ-9 has 9 items, each of which is scored 0,1,2,3, leading to a maximum score of 27. The total scores of 5, 10, 15 and 20 are taken as mild, moderate, moderately severe and severe in terms of the questioner's depressive illness. Cronbach's alpha for PHQ-9 was 0.91. The reliability was further supported by split-half reliability for PHQ-9; part 1 (r = 0.86), part 2 (r = 0.84) and correlation between two halves (r = 0.77), Spearman Brown coefficient was 0.87, and Guttmann split-half coefficient was 0.8.
Generalized Anxiety Disorder 7-item scale (GAD-7) | at Pre-Assessment, after 5 weeks at post-Assessment
  The Generalized Anxiety Disorder 7-item scale (GAD-7) is a widely used self-report screening tool designed to assess the severity of generalized anxiety symptoms. Developed by Spitzer et al. (2006), the scale consists of 7 items, each rated on a 4-point Likert scale ranging from 0 (not at all) to 3 (nearly every day), with total scores ranging from 0 to 21. Higher scores indicate greater levels of anxiety. The GAD-7 has demonstrated high internal consistency, with a Cronbach's alpha of 0.92, and test-retest reliability of 0.83, making it a reliable instrument for both clinical and research use. In the present study, the GAD-7 will be used to measure anxiety symptoms before and after the intervention, allowing evaluation of the impact of Adapted CBT on comorbid anxiety in patients with Major Depressive Disorder.
WHOQOL BREF Scale (WHO; Skevington, Lotfy &Connell, 2004). | at pre-assessment, after 5 weeks at post-assessment
  WHO developed WHOQOL BREF scale. In the current study WHOQOL Brief scale translated by (Ahmad, Hussain, Akhtar & Shah, 2018). The WHOQOL-Brief, still in field trials, is a subset of 26 items taken from the WHOQOL-100. The same steps for the scoring WHOQOL-100 should be followed to achieve scores for the Brief. The four domain scores are scaled in a positive direction with higher scores indicating a higher quality of life. Three items of the Brief must be reversed before scoring.
Mental Help-Seeking Attitudes Scale (MHSAS), | at pre-assessment, after 5 weeks at post-assessment
  The Mental Help-Seeking Attitudes Scale (MHSAS), developed by Hammer, Parent, and Spiker (2018), is a 9-item self-report instrument designed to assess individuals' overall attitudes toward seeking help from mental health professionals. Each item is rated on a 7-point semantic differential scale (e.g., harmful-beneficial, useless-useful), with higher scores indicating more positive attitudes toward mental health help-seeking. The MHSAS has demonstrated strong psychometric properties, including high internal consistency with a Cronbach's alpha of approximately .93, and strong test-retest reliability. The scale has also shown construct validity, being significantly correlated with related variables such as stigma, norms, and intention to seek help.
Motivation and Attitudes Toward Changing Health (MATCH) | at pre-assessment, after 5 weeks at post-assessment
  The Motivation and Attitudes Toward Changing Health (MATCH) scale, developed by Hessler et al. (2018) at the Behavioral Diabetes Institute, is a concise 9-item self-report measure designed to evaluate patients' readiness for health-related behavior change. It includes three subscales: Willingness to Change, Perceived Ability to Change, and Belief that Change is Worthwhile, each containing 3 items. Responses are rated on a 5-point Likert scale, with some items reverse-scored. The MATCH scale has shown acceptable internal consistency, with Cronbach's alpha values ranging from 0.61 to 0.74 across subscales, and has demonstrated good construct validity.
Digit Span Test ( Backward and Forward) | at pre-assessment, after 5 weeks, post-assessment
  The Digit Span Test, a subtest of the Wechsler Adult Intelligence Scale (WAIS), is used to assess attention, concentration, and working memory. It includes two components: Digit Span Forward and Digit Span Backward. In the Forward task, participants repeat a sequence of numbers in the same order as presented, primarily measuring attention span and short-term memory. In the Backward task, participants repeat the numbers in reverse order, assessing working memory and mental manipulation abilities. Typically, performance is higher on the forward span than the backward span due to the increased cognitive demands of the latter. The Digit Span Test has demonstrated adequate internal consistency and reliability, with reported Cronbach's alpha values ranging from .80 to .90, indicating strong psychometric properties for assessing cognitive functioning related to attention and memory.

CONTACTS AND LOCATIONS:
Overall Officials: Qasir Abbas Dr, PhD Clinical Psychology, Principal Investigator — Government College University Faisalabad
Locations (1):
- Government College University Faisalabad, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No